CLINICAL TRIAL: NCT04130672
Title: Hot Nasal Packing With Hot Saline Irrigation for Hemostasis After Adenoidectomy: A Prospective Randomized Controlled Study
Brief Title: Hot Nasal Packing With Hot Saline Irrigation for Hemostasis After Adenoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Mahmut Alper Kanmaz, Assistant Professor, Sanko University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: akanmaz
Record Dates: First submitted 2019-08-19; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Hemostasis After Adenoidectomy
Keywords: Hot tampon; hot saline; adenoidectomy; hemostasis; bleeding control

STUDY DESIGN:
Intervention Model Description: A Prospective Randomized Controlled Study
Who Masked: Investigator
Masking Description: Single blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot saline irrigation (Other): . After adenoidectomy, tonsil tampon at room temperature or 50 ° C was placed in the nasopharynx. Five minutes later, the tampon was removed, and 50 ° C saline irrigation was applied.
  Interventions: Procedure: Hot nasal packing with hot saline irrigation for hemostasis after adenoidectomy
- Cold saline irrigation (Other): . After adenoidectomy, tonsil tampon at room temperature or 22 ° C was placed in the nasopharynx. Five minutes later, the tampon was removed, and 22 ° C saline irrigation was applied.
  Interventions: Procedure: Cold nasal packing with cold saline irrigation for hemostasis after adenoidectomy

INTERVENTIONS:
Procedure: Hot nasal packing with hot saline irrigation for hemostasis after adenoidectomy — After hot packing nasopharyngeal irrigation with 50 C saline
  Arms: Hot saline irrigation
Procedure: Cold nasal packing with cold saline irrigation for hemostasis after adenoidectomy — After cold packing nasopharyngeal irrigation with 22 C saline
  Arms: Cold saline irrigation

SUMMARY:
Objective: This study aimed to investigate the efficacy of hot posterior nasal packing and hot saline irrigation in bleeding control after adenoidectomy.

Methods: 130 patients scheduled for the only adenoidectomy were included, and randomized into two groups at the beginning of the surgical operation. After adenoidectomy, saline impregnated tampon, and saline irrigation at room temperature (22 ° C) was applied to the patients in one group while 50 °C saline impregnated tampon and saline irrigation at the same temperature were applied to the patients in the other group. We record the time for up to 3 minutes after tamponage for bleeding control, bleeding volume, and the amount of bleeding in the nasopharynx

DETAILED DESCRIPTION:
A prospective controlled randomized, single-blind study was designed to investigate the effect of a hot tampon with hot saline irrigation in hemostasis of adenoidectomy. After the parents signed informed consent, the patients under the age of 16 years, who underwent adenoidectomy due to the chronic nasal obstruction, were included in this study. Patients with chronic diseases, patients with bleeding diseases, and patients who had additional procedures were excluded from the study. Among 137 patients who met the inclusion criteria, one hundred and thirty patients agreed to give an informed consent form were included in the study. Under the Declaration of Helsinki, the study protocol was approved by the Clinical Research Ethics Committee (Permit number:5/2019 ).

The patients were divided into 22 ° C and 50 ° C irrigation groups using a computerized random number chart for each working day. To provide blind-evaluation of bleeding by the surgeon, a nurse organized heating the tampon and water, placed both nostrils latex Foley catheters and performed the irrigation processes.

The temperature of the irrigation water and the tampon was adjusted through mixing hot and cold water while immersing a thermometer in the water. The temperature of the irrigation fluid was also controlled every minute to make sure it is a constant value of 50 °C (Fig. 1).

All operations will be performed under general anesthesia and a flexible fiberoptic endoscope carefully assessed adenoid size before the operation with the following grading system: grade 1 (<1/3 of posterior choanae obstructed), grade 2 (1/3-2/3 of posterior choanae obstructed) and grade 3 (>2/3 of posterior choanae obstructed) [13]. Following the patients lay down with Rose's position which their head and neck were extended by placing rolls under the shoulder, the Boyle-Davis mouth retractor was placed, and adenoidectomy was performed via curettes. Complete excision was confirmed by digital palpation and nasopharyngeal mirror. After adenoidectomy, tonsil tampon at room temperature or 50 ° C was placed in the nasopharynx. Five minutes later, the tampon was removed, and 22 ° C or 50 ° C saline irrigation was applied. The scoring system described by Boezaart et al. [14] was adapted to the nasopharynx and using this scoring system and the direct visual observation instead of scoring endoscopy, the nasopharynx was scored and recorded at four different time points: after just tamponing, at the end of one, two and three minutes. The scoring was consisted of following scores: 0=there is no bleeding, 1=accumulation in the nasopharynx is very slow and slightly leak, 2= nasopharynx filling if not aspirated intermittently, 3= blood accumulation in the nasopharynx requiring frequent aspiration, 4= nasopharynx filling if not continuously aspirated, 5= severe bleeding overflowing to the oropharynx. The scoring process was terminated when the washing liquid was clean from bleeding during the irrigation. If this washing time was less than 3 minutes, bleeding scores at remaining time points were also accepted as 0. The irrigation fluids were applied at a rate of about 150 ccs per minute and not exceeding 500 ccs in total. When the irrigation time exceeded 3 minutes, the procedure was stopped to control the bleeding through bipolar cauterization, and the irrigation was continued with saline at the same temperature. The amount of bleeding was determined by removing the volume of irrigation fluid from the volume of the material accumulated in the aspirator chamber. The bleeding site and residual adenoid were detected by the nasopharyngeal mirror.

ELIGIBILITY:
Inclusion Criteria:

The patients who underwent adenoidectomy

Exclusion Criteria:

* Patients with chronic diseases
* Patients with bleeding diseases

Ages: 18 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
Bleeding time | through bleeding control , an average of 5 minutes
  Depanding on which type of saline irrigation and packing used after adenoidectomy

SECONDARY OUTCOMES:
Bleeding amount | through bleeding control , an average of 5 minutes
  Depanding on which type of saline irrigation and packing used after adenoidectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmut Alper Kanmaz, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
ıf anyone requires the patient's data